CLINICAL TRIAL: NCT01678105
Title: A Phase II Study of DOVitinib in REcurrent and/or Metastatic Adenoid Cystic Carcinoma of the Salivary Glands (DOVE)
Brief Title: A Phase II Study of Dovitinib in Recurrent and/or Metastatic Adenoid Cystic Carcinoma of the Salivary Glands
Acronym: DOVE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ontario Clinical Oncology Group (OCOG) (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OCOG-2012-DOVE
Record Dates: First submitted 2012-08-23; First posted 2012-09-03 (Estimated); Last update posted 2015-09-17 (Estimated); Status verified 2015-09

CONDITIONS: Recurrent Adenoid Cystic Carcinoma of the Salivary Glands; Metastatic Adenoid Cystic Carcinoma of the Salivary Glands; Salivary Gland Cancers; ACC
Keywords: Recurrent Adenoid Cystic Carcinoma of the Salivary Glands; Metastatic Adenoid Cystic Carcinoma of the Salivary Glands; Salivary Gland Cancers; ACC; Dovitinib; TKI258; RTK Inhibitor
MeSH Terms: conditions — Salivary Gland Neoplasms | interventions — 4-amino-5-fluoro-3-(5-(4-methylpiperazin-1-yl)-1H-benzimidazol-2-yl)quinolin-2(1H)-one

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dovitinib (Experimental): Dovitinib 500 mg PO OD (5 days on, 2 days off); Each cycle = 28 days
  Interventions: Drug: Dovitinib

INTERVENTIONS:
Drug: Dovitinib — Treatment continued until Disease Progression, Toxicity, or patient withdrawal
  Other Names: TKI258; RTK Inhibitor

SUMMARY:
This is a non-randomized, phase II, open label study of dovitinib in patients with progressive, recurrent and/or metastatic adenoid cystic carcinoma (ACC). The primary purpose of this study is to assess the anti-cancer effects of dovitinib in this population in order to evaluate whether dovitinib is worthy of further study in patients with progressive ACC.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed ACC of major or minor salivary glands.
* Recurrent and/or metastatic disease deemed progressive that is not amenable to surgery or curative radiotherapy.
* Measurable disease according to the Response Evaluation Criteria in Solid Tumors (RECIST, version 1.1), defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter in the plane of measurement is to be recorded) with a minimum size of:

  * > 10 mm by CT scan (CT scan slice thickness no greater than 5 mm).
  * > 10 mm caliper measurement by clinical exam (lesion which cannot be accurately measured with calipers should be recorded as non-measurable).
  * > 20 mm by chest X-ray Malignant lymph nodes: To be considered pathologically enlarged and measurable, a lymph node must be >15mm in short axis when assessed by CT scan (CT scan slice thickness recommended to be no greater than 5 mm).
* Progressive disease, defined as one of the following occurring within 12 months of study entry:

  i) at least a 10% increase in radiologically or clinically measurable disease; ii) appearance of one or more new lesions, or iii) deterioration in clinical status.

Exclusion Criteria:

* Less than 18 years of age.
* Life expectancy < 12 weeks.
* ECOG performance status > 2.
* Known brain metastases.
* Treatment with chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Major surgery within 4 weeks prior to entering the study.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to dovitinib.
* Taking medications that are potent CYP3A4 inducers or inhibitors (dovitinib is metabolized primarily by the CYP3A4 liver enzyme, every effort should be made to switch patients taking such agents or substances to other medications).
* History of cardiac dysfunction with an ECHO or MUGA scan outside the institutional range of normal.
* QTc prolongation (defined as a QTc interval > 500 msec) or other significant ECG abnormalities.
* Poorly controlled hypertension (systolic blood pressure of ≥ 140 mmHg or diastolic blood pressure of ≥ 90 mmHg).
* Any abnormal organ and marrow function as defined below:

  * Leukocytes <3,000/microL
  * Absolute neutrophil count <1,500/microL
  * Platelets <100,000/microL
  * Total bilirubin >1.5X institutional upper limit of normal (ULN)
  * AST(SGOT) / ALT(SGPT) >2.5X institutional ULN
  * Amylase/lipase outside normal institutional limits
  * Serum creatinine >1.5X ULN
  * Creatinine clearance <60mL/min/1.73 m2 for patients with creatinine levels above institutional normal
* Required use of therapeutic doses of coumarin-derivative anticoagulants such as warfarin, although doses of up to 2mg daily are permitted for prophylaxis of thrombosis. Note: Low molecular weight heparin is permitted provided the patient's PT INR is ≤ 1.5.
* Pre-existing condition (e.g., gastrointestinal tract disease), resulting in an inability to take oral medication or a requirement for IV alimentation, prior surgical procedures affecting absorption, or active peptic ulcer disease that impairs their ability to swallow and retain dovitinib tablets.
* Pre-existing thyroid abnormality with an inability to maintain thyroid function in the normal range with medication.
* Any of the following conditions:

  * Serious or non-healing wound, ulcer, or bone fracture,
  * History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 28 days of treatment,
  * History of cerebrovascular accident (CVA) or transient ischemic attack (TIA) within 12 months prior to study entry,
  * History of pulmonary embolism within the past 12 months,
  * History of myocardial infarction, cardiac arrhythmia, stable/unstable angina, symptomatic congestive heart failure, or coronary/peripheral artery bypass graft or stenting within 12 months prior to study entry,
  * NYHA Class III or IV heart failure as defined by the NYHA functional classification system.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infections, HIV-positive patients on combination antiretroviral therapy.
* Pregnant or lactating women.
* Psychiatric illness/social situations that would limit compliance with study requirements.
* Receiving any other investigational agent(s).
* Inability to understand or unable to provide written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2012-11; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Clinical Benefit Rate | 2 years
  The primary outcome measure is the clinical benefit rate, defined as an objective response (complete [CR] or partial [PR]) or stable disease [SD] of ≥6 months duration according to the RECIST version 1.1 criteria.

SECONDARY OUTCOMES:
Progression Free Survival | From the date the patient first receives study medication to the date of death or date of progression according to RECIST or symptomatic deterioration; estimated to be after 12 weeks of treatment
Overall Survival | From the date the patient first receives study medication to the date of death; patients will be followed up for survival for up to 2 years after disease progression
Safety and tolerability | From the date the patient first receives study medication to the date the patient completes the study; patients will be followed up for survival for up to 2 years after disease progression
  Patients will be evaluated for toxicity. Frequency and severity of adverse events will be tabulated using counts and proportions detailing frequently occuring, serious and severe events of interest.

CONTACTS AND LOCATIONS:
Overall Officials: Sebastien Hotte, MD, Principal Investigator — Juravinski Cancer Centre; Mark Levine, MD, Study Director — Ontario Clinical Oncology Group (OCOG); Greg Pond, PhD, Principal Investigator — Ontario Clinical Oncology Group (OCOG)
Locations (4):
- Canada (4):
  - Tom Baker Cancer Centre, Calgary, Ontario
  - Juravinski Cancer Centre, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - Ottawa Hospital Regional Cancer Centre, Ottawa, Ontario